CLINICAL TRIAL: NCT05207865
Title: A Phase 4, Open-label Study to Evaluate the Safety and Tolerability of Daily Dosing of Rimegepant in Episodic Migraine Prevention
Brief Title: Safety and Tolerability Study of Daily Dosing Rimegepant in Episodic Migraine Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV3000-405; C4951011 (Other: Alias Study Number)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Migraine; Episodic Migraine; Phonophobia; Photophobia
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rimegepant (Experimental): rimegepant 75 mg ODT daily
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — rimegepant ODT 75mg daily
  Other Names: BHV-3000

SUMMARY:
The purpose of this study is to further evaluate the long-term safety and tolerability of daily dosing of rimegepant for the prevention of episodic migraine.

DETAILED DESCRIPTION:
This is a post marketing required study being conducted to further evaluate the long-term safety and tolerability of a more frequent daily dosing regimen of rimegepant for the prevention of episodic migraine.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has at least 1 year history of episodic migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:
* Age of onset of migraines prior to 50 years of age
* Migraine attacks, on average, lasting 4 -72 hours if untreated
* Per subject report, 4-14 migraine attacks per month within the last 3 months prior to the Screening Visit (month is defined as 4 weeks for the purpose of this protocol)
* Subjects ≥ 18 years

Key Exclusion Criteria:

* Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with myocardial infarction (MI), acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months (24 weeks) prior to the Screening Visit.
* Uncontrolled hypertension (high blood pressure) or uncontrolled diabetes.
* The subject has a history or current evidence of any unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known or suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the study
* History of use of opioid- or barbiturate- (e.g. butalbital) containing medication for 4 or more days per month during the 3 months (12 weeks) prior to the Screening Visit
* WOCBP who are unwilling or unable to use an acceptable contraceptive method or abstinence to avoid pregnancy for the entire study and for 28 days after the last dose of study drug
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test at screening or prior to study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Velocity Clinical Research - North Hollywood, North Hollywood, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Phoenix Medical Research, LLC, Miami, Florida
  - The Headache Clinic, Alexandria, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - CVS HealthHub - East Brunswick, East Brunswick, New Jersey
  - CVS HealthHub - Lawrenceville, Lawrenceville, New Jersey
  - CVS HealthHUB - Runnemede, Runnemede, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Velocity Clinical Research, Cincinnati, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Clinical Research Philadelphia, LLC, Philadelphia, Pennsylvania
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - VIP Trails, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Antinew J, Fountaine RJ, Loprinzo V, Straghan E, Dubrovin S, DeBesi P, Vatakis N, Fullerton T. A phase 4, 24-week, open-label study to evaluate the safety and tolerability of once-daily dosing of 75 mg rimegepant for episodic migraine prevention. J Headache Pain. 2025 Dec 9;27(1):17. doi: 10.1186/s10194-025-02225-7. PMID 41366286
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-405

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 441 enrolled participants, only 250 received study treatment; 184 participants failed screening, 6 participants were lost to follow-up and 1 participant withdrew consent.
Groups:
- Rimegepant: Participants received a single dose of Rimegepant 75 milligrams (mg) orally disintegrating tablet (ODT) daily for 24 weeks during the open-label treatment phase.
Period: Open-Label Treatment Phase
Arm/Group | Rimegepant
Started | 250
Completed | 187
Not Completed | 63
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 8
Not completed — Non-compliance | 3
Not completed — Other | 17
Not completed — Physician Decision | 2
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 1
Not completed — Protocol-specified withdrawal criterion met | 14
Not completed — Withdrawal by Subject | 10
Period: Follow-up Phase
Arm/Group | Rimegepant
Started (Participants who took study drug whose last contact date is in the follow-up analysis period.) | 235
Completed | 220
Not Completed | 15
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance | 1
Not completed — Not reported | 2
Not completed — Not collected | 11

BASELINE CHARACTERISTICS:
Groups:
- Rimegepant: Participants received a single dose of Rimegepant 75 mg ODT daily for 24 weeks during the open-label treatment phase.
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35
  Not Hispanic or Latino | 215
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 216
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-Treatment Adverse Events (AEs) (Frequency >=5%) According to Intensity
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered an investigational (medicinal) product and did not necessarily have causal relationship with treatment. On-treatment AEs were those AEs which occurred after the study treatment start date until 7 days after last dose of study treatment. AEs were classified according to intensity as: mild: transient and required minimal treatment or therapeutic intervention, event did not interfere with usual activities of daily living; moderate: alleviated with additional specific therapeutic intervention, event interfered with activities of daily living, causing discomfort; severe: interrupted activities of daily living, affected clinical status, or required intensive treatment. AEs occurring in >=5% participants are reported in this OM.
Time Frame: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks)
Population: Safety analysis set included participants in the enrolled analysis set who took greater than or equal to (>=) 1 dose of study drug (rimegepant), i.e., nonmissing study drug start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Participants
  Mild | 33
  Moderate | 17
  Moderate or severe | 17

2. Primary Outcome: Number of Participants With On-Treatment Serious Adverse Events (SAEs)
Description: An SAE was any event that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; was persistent or caused significant disability/incapacity or congenital anomaly/birth defect in the offspring of a participant who received Rimegepant, or other important medical events. On-treatment AEs were those AEs which occurred after the study treatment start date until 7 days after last dose of study treatment.
Time Frame: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks)
Population: Safety analysis set included participants in the enrolled analysis set who took >= 1 dose of study drug (rimegepant), i.e., nonmissing study drug start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Participants | 0

3. Primary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered an investigational (medicinal) product and did not necessarily have causal relationship with treatment. Number of participants with AEs leading to study drug discontinuations are reported in this outcome measure.
Time Frame: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Participants | 7

4. Primary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities On-Treatment Using Common Technical Criteria for Adverse Events- Division of Acquired Immune Deficiency Syndrome (CTCAE/DAIDS) Toxicity Grading Scale
Description: The following laboratory parameters were assessed: eosinophils, hemoglobin low and high, leukocytes low, lymphocytes low and high, neutrophils, platelets, alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, calcium low and high, cholesterol, creatine kinase, creatinine, glomerular filtration rate estimated, glucose low and high, lactate dehydrogenase, low-density lipoprotein (LDL) cholesterol, LDL cholesterol fasting and not fasting, potassium low and high, sodium low and high, triglycerides, triglycerides fasting and not fasting, uric acid, urine glucose and urine protein. Laboratory abnormalities were graded according to NCI CTCAE v5.0; where grade 3=severe and grade 4=life-threatening except for glucose, LDL cholesterol, and urinalysis where DAIDS v2.1 was used. (grade 3= severe and grade 4= life-threatening).
Time Frame: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks)
Population: Safety analysis set included participants in the enrolled analysis set who took >= 1 dose of study drug (rimegepant), i.e., nonmissing study drug start date. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row and "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Participants
  Eosinophils: number analyzed (Participants) | 237
  Eosinophils | 0
  Hemoglobin, low: number analyzed (Participants) | 237
  Hemoglobin, low | 0
  Hemoglobin, high: number analyzed (Participants) | 237
  Hemoglobin, high | 0
  Leukocytes, low: number analyzed (Participants) | 237
  Leukocytes, low | 0
  Lymphocytes, low: number analyzed (Participants) | 237
  Lymphocytes, low | 1
  Lymphocytes, high: number analyzed (Participants) | 237
  Lymphocytes, high | 0
  Neutrophils: number analyzed (Participants) | 237
  Neutrophils | 0
  Platelets: number analyzed (Participants) | 237
  Platelets | 0
  Alanine Aminotransferase: number analyzed (Participants) | 237
  Alanine Aminotransferase | 0
  Albumin: number analyzed (Participants) | 237
  Albumin | 0
  Alkaline Phosphatase: number analyzed (Participants) | 237
  Alkaline Phosphatase | 0
  Aspartate Aminotransferase: number analyzed (Participants) | 237
  Aspartate Aminotransferase | 0
  Bicarbonate: number analyzed (Participants) | 237
  Bicarbonate | 0
  Bilirubin: number analyzed (Participants) | 237
  Bilirubin | 0
  Calcium, low: number analyzed (Participants) | 237
  Calcium, low | 0
  Calcium, high: number analyzed (Participants) | 237
  Calcium, high | 0
  Cholesterol: number analyzed (Participants) | 225
  Cholesterol | 0
  Creatine Kinase: number analyzed (Participants) | 237
  Creatine Kinase | 9
  Creatinine: number analyzed (Participants) | 237
  Creatinine | 0
  Glomerular Filtration Rate, Estimated: number analyzed (Participants) | 237
  Glomerular Filtration Rate, Estimated | 0
  Glucose, low: number analyzed (Participants) | 236
  Glucose, low | 1
  Glucose, high: number analyzed (Participants) | 236
  Glucose, high | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 236
  Lactate Dehydrogenase | 0
  LDL Cholesterol: number analyzed (Participants) | 225
  LDL Cholesterol | 22
  LDL Cholesterol, fasting: number analyzed (Participants) | 150
  LDL Cholesterol, fasting | 14
  LDL Cholesterol, not fasting: number analyzed (Participants) | 88
  LDL Cholesterol, not fasting | 9
  Potassium, low: number analyzed (Participants) | 236
  Potassium, low | 0
  Potassium, high: number analyzed (Participants) | 236
  Potassium, high | 3
  Sodium, low: number analyzed (Participants) | 237
  Sodium, low | 0
  Sodium, high: number analyzed (Participants) | 237
  Sodium, high | 0
  Triglycerides: number analyzed (Participants) | 225
  Triglycerides | 2
  Triglycerides, fasting: number analyzed (Participants) | 150
  Triglycerides, fasting | 2
  Triglycerides, not fasting: number analyzed (Participants) | 88
  Triglycerides, not fasting | 0
  Uric Acid: number analyzed (Participants) | 237
  Uric Acid | 0
  Urine Glucose: number analyzed (Participants) | 209
  Urine Glucose | 1
  Urine Protein: number analyzed (Participants) | 209
  Urine Protein | 0

5. Primary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities On-Treatment Using Food and Drug Administration (FDA) Toxicity Grading Scale
Description: The following laboratory parameters were assessed: eosinophils, hemoglobin, leukocytes low, lymphocytes low and high, neutrophils, platelets, alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, blood urine nitrogen, calcium low and high, cholesterol, creatine, glucose low and high, potassium low and high, protein, sodium low and high, urine glucose and urine protein. Laboratory abnormality events were graded according to FDA toxicity grading scale (grade 3= severe and grade 4= life-threatening).
Time Frame: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant
Number analyzed (Participants) | 250
Participants
  Eosinophils: number analyzed (Participants) | 237
  Eosinophils | 0
  Hemoglobin: number analyzed (Participants) | 237
  Hemoglobin | 4
  Leukocytes, low: number analyzed (Participants) | 237
  Leukocytes, low | 0
  Leukocytes, high: number analyzed (Participants) | 237
  Leukocytes, high | 0
  Lymphocytes: number analyzed (Participants) | 237
  Lymphocytes | 1
  Neutrophils: number analyzed (Participants) | 237
  Neutrophils | 0
  Platelets: number analyzed (Participants) | 237
  Platelets | 0
  Alanine Aminotransferase: number analyzed (Participants) | 237
  Alanine Aminotransferase | 0
  Albumin: number analyzed (Participants) | 237
  Albumin | 0
  Alkaline Phosphatase: number analyzed (Participants) | 237
  Alkaline Phosphatase | 0
  Aspartate Aminotransferase: number analyzed (Participants) | 237
  Aspartate Aminotransferase | 0
  Bilirubin: number analyzed (Participants) | 237
  Bilirubin | 1
  Blood Urine Nitrogen: number analyzed (Participants) | 237
  Blood Urine Nitrogen | 1
  Calcium, low: number analyzed (Participants) | 237
  Calcium, low | 0
  Calcium, high: number analyzed (Participants) | 237
  Calcium, high | 0
  Cholesterol: number analyzed (Participants) | 225
  Cholesterol | 54
  Creatinine: number analyzed (Participants) | 237
  Creatinine | 0
  Glucose, low: number analyzed (Participants) | 236
  Glucose, low | 4
  Glucose, high: number analyzed (Participants) | 236
  Glucose, high | 19
  Potassium, low: number analyzed (Participants) | 236
  Potassium, low | 0
  Potassium, high: number analyzed (Participants) | 236
  Potassium, high | 10
  Protein: number analyzed (Participants) | 237
  Protein | 1
  Sodium, low: number analyzed (Participants) | 237
  Sodium, low | 0
  Sodium, high: number analyzed (Participants) | 237
  Sodium, high | 6
  Urine Glucose: number analyzed (Participants) | 209
  Urine Glucose | 1
  Urine Protein: number analyzed (Participants) | 209
  Urine Protein | 0

ADVERSE EVENTS:
Time Frame: For On-treatment period: From start of study treatment (Day 1) up to 7 days after the last dose of study treatment (Up to 25 weeks); For Follow-up period- from 2 weeks after last dose of study treatment up to 8 weeks after last dose of study treatment
Description: Safety analysis set included participants in the enrolled analysis set who took >= 1 dose of study drug (rimegepant), i.e., nonmissing study drug start date.
Groups:
- Rimegepant (On-treatment Period): Participants received a single dose of Rimegepant 75 mg ODT daily for 24 weeks during the open-label treatment phase.
- Rimegepant (Follow-up Period): Participants were followed up from 2 weeks after last dose of study treatment up to 8 weeks after last dose of study treatment.
Arm/Group | Rimegepant (On-treatment Period) | Rimegepant (Follow-up Period)
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/235
Serious Adverse Events (participants affected / at risk) | 0/250 | 2/235
Other Adverse Events (participants affected / at risk) | 48/250 | 2/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant (On-treatment Period) (N=250) | Rimegepant (Follow-up Period) (N=235)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant (On-treatment Period) (N=250) | Rimegepant (Follow-up Period) (N=235)
Nasopharyngitis (Infections and infestations) | 23 | 1
COVID-19 (Infections and infestations) | 16 | 0
Nausea (Gastrointestinal disorders) | 15 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT05207865/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT05207865/SAP_001.pdf